CLINICAL TRIAL: NCT03526822
Title: Prospective Cohort of Patients With Newly Diagnosed Glioblastoma: Analysis of MMP2 and MMP9 Expression and Correlation to Neuro-imaging Features.
Acronym: MM-Predict
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-56; 2018-A00740-55 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with newly diagnosed glioblastoma (Experimental)
  Interventions: Biological: Blood sample; Biological: Tumor sample

INTERVENTIONS:
Biological: Blood sample — Five blood sample in pre-, post-operative period, before radiotherapy, before adjuvant temozolomide and at relapse in newly diagnosed glioblastoma
Biological: Tumor sample — One tumor sample in operative period

SUMMARY:
Glioblastoma is the most frequent and aggressive primary brain tumor in adults. A team recently showed that baseline plasma levels of matrix metalloproteinase-2 (MMP2) and matrix metalloproteinase-9 (MMP9) were correlated to bevacizumab activity in patients with recurrent glioblastoma. To date, the biological rationale of this results remains unknown but MMP2 could be involved in classical angiogenesis while MMP9 could promote vasculogenesis.

The objectives are to correlate the plasma levels of MMP2 and MMP9 to their Ribonucleic acid (RNA) and protein tissue expression, activity and to patient neuro-imaging features. To analyze the changes of MMP2 and MMP9 plasma levels during peri-operative period and after radio-chemotherapy.

Methods: Plasmatic levels of MMP2, MMP9, vascular endothelial growth factor-A (VEGFA), vascular endothelial growth factor-R2 (VEGFR2), stromal cell-derived factor 1 (SDF1) and chemokine receptor-4 (CXCR4) will be analyzed by enzyme-linked immunosorbent assay (ELISA) in pre-, post-operative period, before radiotherapy, before adjuvant temozolomide and at relapse in newly diagnosed glioblastoma. RNA expression of these factors will be analyzed by reverse transcription-Polymerase chain reaction (RT-qPCR) on frozen tumor samples, whereas protein expression will be analyzed by ELISA and immunohistochemistry. Enzymatic activity of MMP2 and MMP9 will be analyzed by zymography. Tumor volume, infiltration and perfusion degrees will be analyzed on Magnetic Resonance Imaging (MRI) performed before and after surgery and before adjuvant temozolomide. Neuro-imaging characteristics will be correlated to plasma and tissue expressions of these factors.

The expected results are to better define the expression profile of MMP2, MMP9 and the change in their plasma level during treatment, a prerequisite for their clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged 18 years or over
* Imaging suggestive of glioblastoma
* Patient eligible for excision surgery (partial, subtotal or macroscopically complete)
* Candidate for concomitant and adjuvant radiotherapy chemotherapy (Stupp protocol)
* Patient having signed an informed consent
* Patient having undergone a preoperative MRI

Exclusion Criteria:

* Existence of a contraindication to the MRI
* Nonoperable lesion
* History of radiotherapy and / or chemotherapy for this lesion
* Scalability of a low grade lesion
* Person in emergency situation, a legal person of legal age (guardianship, guardianship or legal guardianship), or unable to express his or her consent
* No affiliation to a social security scheme (beneficiary or beneficiary)
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
correlate the plasma levels of MMP2 and MMP9 to their RNA and protein tissue expression by ELISA | 18 months
  identify potential temporal variations of these markers

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France